CLINICAL TRIAL: NCT01792661
Title: Navigating the Challenges of Chronic Kidney Disease
Acronym: CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 12-072; R34DK094112-01 (NIH)
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Electronic Health Record; Personal Health Record; Chronic Kidney Disease registry; Glomerular Filtration Rate; Patient Navigator
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Patient Navigation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MyChart (Active Comparator): The control group receives standard Cleveland Clinic care and has access to MyChart which is the standard Cleveland Clinic electronic PHR.
  Interventions: Other: MyChart
- Enhanced MyChart (Active Comparator): The enhanced PHR functionality adds the ability to securely receive and review CKD-education related messages to the existing features available to all PHR users. The CKD-educational related messages can be automatically delivered at pre-defined intervals and customized for each individual patient at their discretion and convenience.
  Interventions: Other: Enhanced MyChart
- Patient Navigator (Active Comparator): A tracking log is kept by the Patient Navigator of each interaction regarding type of encounter, length of encounter, barriers addressed, and actions that occurred, adapting what is in use for the NIH-funded Patient Navigator program.
  Interventions: Other: Patient Navigator; Other: MyChart
- Patient Navigator and Enhanced MyChart (Active Comparator): Combines patient self empowerment, regarding their CKD, with the Enhanced MyChart along with the aid and direction of a Patient Navigator.
  Interventions: Other: Enhanced MyChart; Other: Patient Navigator

INTERVENTIONS:
Other: Enhanced MyChart — Subjects randomized into the MyChart receive an additional site on their MyChart containing 35 extra educational links specific to CKD, targetting care for stage 3b and stage 4 patients.
  Other Names: CKD Enhanced PHR
  Arms: Enhanced MyChart; Patient Navigator and Enhanced MyChart
Other: Patient Navigator — The Patient Navigator aids subjects in education of their CKD, timely scheduling of appointments, plus determining and overcoming barriers to their CKD health care. The Patient Navigator's job is not part of routine medical care.
  Arms: Patient Navigator; Patient Navigator and Enhanced MyChart
Other: MyChart — Sign-up to MyChart is optional for Cleveland Clinic patients. Subjects enrolled into the study are signed-up for MyChart (if not already signed-up) during the consenting process.
  Arms: MyChart; Patient Navigator

SUMMARY:
The study's purpose is to address the challenges of providing stage-appropriate chronic kidney disease (CKD) education and care by developing innovative programs using a CKD Patient Navigator system and an EHR (electronic health record)-based enhanced electronic communication system specific for a CKD patient and her/his physicians/caregivers. The investigators plan a randomized controlled trial of these innovations to examine the utility and effectiveness of these special interventions.

The investigators' CKD registry aids in identifying patients for recruitment for the randomized control trial. Patients are randomized into one of four groups. The four groups are: 1) the control group using MyChart; 2) an enhanced personal health record (PHR) included in MyChart consisting of 35 websites chosen to disseminate CKD stage-specific goals of care and CKD education; 3) the patient navigator, a lay professional trained in the specifics of chronic kidney disease navigation with a focus on the needs of their patients based on the National Kidney Foundation Disease Outcomes Quality Initiative; 4) the patient navigator combined with the enhanced MyChart.

The investigators hypothesize that a CKD Patient Navigator program will develop a more prepared, proactive patient-caregiver team than usual care; the enhanced PHR will produce a more informed, engaged patient than usual care; the CKD Patient Navigator arm and enhanced PHR will demonstrate a slower rate of decline in eGFR (glomerular filtration rate) than usual care.

The results of this study will lay the foundation for a larger multi-center national clinical trial that will build upon the feasibility and knowledge gained from this planning grant.

DETAILED DESCRIPTION:
The overall goal of this research is to assess the effects of innovative interventions for CKD on the decline in renal function among patients with CKD stages 3b or 4. First, a CKD Patient Navigator program was created, adapted from the use of Patient Navigators successfully in oncology. Second, an enhanced PHR was developed that uses electronic communication to disseminate CKD stage-specific goals of care and CKD education. Third, a randomized controlled trial is being conducted using a factorial design to investigate the clinical impact and cost-effectiveness of the two interventions - a CKD Patient Navigator and enhanced PHR compared to usual care for CKD Stage 3b/4 patients.

As a conceptual framework for the proposed study, the investigators are using the Chronic Care Model developed by Edward H. Wagner, M.D., Director of The MacColl Institute for Healthcare Innovation, Director of The Robert Wood Johnson Foundation national program "Improving Chronic Illness Care" and Senior Investigator at the Group Health Research Institute in Seattle. The model emphasizes a synergy between community, the health care system, technology and personal interactions to achieve optimal functional and clinical outcomes among people with chronic diseases. It has been adopted by the National Kidney Disease Education Program (NKDEP) to achieve many of their goals related to kidney disease.

With the help of the CKD registry, the investigators are recruiting patients from outpatient clinics at main campus and family health centers located in the surrounding Cleveland area. Patients are being recruited by a trained study coordinator. All patients are informed about study procedures and the purpose of the research, verbally and in a written informed consent document, two copies of which must be signed by both the patient and the study coordinator before enrollment. Upon enrollment, the patients will be provided with a $25 stipend.

The investigators identify from the CKD Registry and recruit eligible patients with CKD stage 3b (eGFR 30-44 ml/min/1.73 m2) or Stage 4 (eGFR 15-29 ml/min/1.73 m2) who meet the inclusion/exclusion criteria. The majority of data comes from the EHR derived CKD registry. The investigators obtain baseline demographic characteristics (age, gender, and race), comorbidities, and medication use, smoking status at the baseline visit. Further, CKD stage specific laboratory data will be collected routinely i.e., whether a laboratory parameter was measured or not and if measured, whether the laboratory measures and blood pressure are under the target limits. Details about nephrology, vascular access, and transplant referrals are obtained at baseline visit. The primary outcome of the study will be change in eGFR over the two-year study period.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* English speaking
* eGFR 15-45 ml/min
* patients residing in North East Ohio

Exclusion Criteria:

* mentally incompetent
* cancer
* terminal illness
* patients on dialysis
* patients who have had renal transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2012-02; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in Renal Function | baseline and 1 year
  CKD stage specific laboratory data is being collected quarterly. Most of the data will come from the CKD registry, supplemented by the data collection system from the EHR set up by the Cleveland Clinic Department of Quantitative Health Sciences (QHS).
  Lab and urine measures are: eGFR, urine albumin to creatinine ratio, parathyroid hormone, 25-OH vitamin D, low density lipoprotein, hemoglobin, calcium and phosphorus.
  Clinical targets are: blood pressure, LDL, 25-OH Vitaming D. Preparation for possible transition to End Stage Renal Disease (ESRD): Nephrology referral, vascular access referral, transplant referral.
  Whether renoprotective medications are prescribed, such as ACEi and ARB.

SECONDARY OUTCOMES:
CKD Knowledge and Awareness | baseline and 1 year
  CKD education is being measured with electronic clicks the number of times NKDEP patient education materials are accessed through Enhanced MyChart, NKF pre-ESRD curriculum.
  Similarly, the frequency of MyChart access of laboratory results and appointments specific to CKD awareness, Nephrology, CKD Clinic, Primary Care Physician, is being measured.
  Nutrition is also being similarly measured; NKDEP nutrition patient education materials, nutrition referral.
  Patient Navigator contact frequency and subsequent patient follow-up of laboratory work and medical appointments are the indicators of patient willingness to increase their CKD knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Nally, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Navaneethan SD, Jolly SE, Schold JD, Arrigain S, Saupe W, Sharp J, Lyons J, Simon JF, Schreiber MJ Jr, Jain A, Nally JV Jr. Development and validation of an electronic health record-based chronic kidney disease registry. Clin J Am Soc Nephrol. 2011 Jan;6(1):40-9. doi: 10.2215/CJN.04230510. Epub 2010 Nov 4. PMID 21051745
- [Background] Navaneethan SD, Kandula P, Jeevanantham V, Nally JV Jr, Liebman SE. Referral patterns of primary care physicians for chronic kidney disease in general population and geriatric patients. Clin Nephrol. 2010 Apr;73(4):260-7. doi: 10.5414/cnp73260. PMID 20353733
- [Background] Jolly SE, Burrows NR, Chen SC, Li S, Jurkovitz CT, Narva AS, Norris KC, Shlipak MG. Racial and ethnic differences in albuminuria in individuals with estimated GFR greater than 60 mL/min/1.73 m(2): results from the Kidney Early Evaluation Program (KEEP). Am J Kidney Dis. 2010 Mar;55(3 Suppl 2):S15-22. doi: 10.1053/j.ajkd.2009.09.034. PMID 20172444
- [Background] Tonelli M, Muntner P, Lloyd A, Manns BJ, James MT, Klarenbach S, Quinn RR, Wiebe N, Hemmelgarn BR; Alberta Kidney Disease Network. Using proteinuria and estimated glomerular filtration rate to classify risk in patients with chronic kidney disease: a cohort study. Ann Intern Med. 2011 Jan 4;154(1):12-21. doi: 10.7326/0003-4819-154-1-201101040-00003. PMID 21200034
- [Background] Chronic Kidney Disease Prognosis Consortium; Matsushita K, van der Velde M, Astor BC, Woodward M, Levey AS, de Jong PE, Coresh J, Gansevoort RT. Association of estimated glomerular filtration rate and albuminuria with all-cause and cardiovascular mortality in general population cohorts: a collaborative meta-analysis. Lancet. 2010 Jun 12;375(9731):2073-81. doi: 10.1016/S0140-6736(10)60674-5. Epub 2010 May 17. PMID 20483451
- [Background] Freeman HP. Patient navigation: a community centered approach to reducing cancer mortality. J Cancer Educ. 2006 Spring;21(1 Suppl):S11-4. doi: 10.1207/s15430154jce2101s_4. PMID 17020496
- [Background] Freund KM. Patient navigation: the promise to reduce health disparities. J Gen Intern Med. 2011 Feb;26(2):110-2. doi: 10.1007/s11606-010-1593-5. No abstract available. PMID 21161422